CLINICAL TRIAL: NCT06431958
Title: Droplet Digital PCR and PCR-free BIOSensors for the Detection of Resistance-associated SNPs in Pneumocystis Jirovecii
Acronym: DDBIOS
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0085 - DDBIOS
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-04

CONDITIONS: Pneumocystis Pneumonia
Keywords: Pneumocystis jirovecii; mutant; anti-microbial resistance; DHPS; DHFR; Cytochrome b; IMPDH
MeSH Terms: conditions — Pneumonia, Pneumocystis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of the proposed research is to identify Pneumocystis jirovecii mutant strains on 4 genes encoding therapeutic targets such as dihydropteroate synthase (DHPS), dihydrofolate reductase (DHFR), cytochrome b (CYB), inosine-5'-monophosphate dehydrogenase (IMPDH) and therefore to assess the prevalence of potentially resistant strains in patients infected with P. jirovecii.

DETAILED DESCRIPTION:
Pneumocystis jirovecii (P. jirovecii) is an opportunistic pathogenic fungus responsible for pulmonary infection or Pneumocystis pneumonia (PCP) in immunocompromised patients. There is currently no system for its in vitro culture. The diagnostic methods used are mainly based on molecular biology techniques which also allow the detection and analysis of single nucleotide polymorphisms (SNPs), particularly at the level of genes coding for the targets of molecules widely used in the prevention and treatment of PCP. These SNPs may represent missense mutations potentially associated with treatment resistance. They may result from exposure of patients to these treatments before the development of P. jirovecii infection. However, data concerning the prevalence of these mutations remains scarce, particularly in France. Methods for detecting these mutations based on PCR followed by DNA sequencing have limitations in terms of sensitivity. The evaluation of new, more sensitive and rapid tools for the detection and characterization of pathogens in this context is necessary.

The main objective of the proposed research is to identify P. jirovecii mutant strains on 4 genes encoding therapeutic targets such as dihydropteroate synthase (DHPS), dihydrofolate reductase (DHFR), cytochrome b (CYB), inosine-5'-monophosphate dehydrogenase (IMPDH) and therefore to assess the prevalence of potentially resistant strains in patients infected with P. jirovecii.

The secondary objectives are:

* to determine the factors associated (e.g. exposure to treatments) with mutant P. jirovecii strains
* to determine the impact of mutations on the effectiveness of anti-Pneumocystis treatment (e.g. favorable vs. unfavorable evolution of the infection)
* to evaluate two methods - digital droplet PCR and biosensors without PCR - for the detection and characterization of mutations associated with resistance in Pneumocystis jirovecii

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom P. jirovecii was detected in a pulmonary sample (bronchoalveolar lavage, sputum, bronchial aspiration, oropharyngeal rinse, nasopharyngeal sample)
* No opposition
* Patient affiliated to a social security system

Exclusion Criteria:

* Patients under legal protection (guardianship, curatorship)
* Refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in whom P. jirovecii was detected in a pulmonary sample (bronchoalveolar lavage, sputum, bronchial aspiration, oropharyngeal rinse, nasopharyngeal sample) can be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of specific strains of Pneumocystis jirovecii potentially resistant to treatments in patients infected with this fungus | at inclusion
  Four genes encoding therapeutic targets such as dihydropteroate synthase (DHPS), dihydrofolate reductase (DHFR), cytochrome b (CYB), inosine-5'-monophosphate dehydrogenase (IMPDH) will be amplified and sequenced to detect single nucleotide polymorphisms (Single Nucleotide Polymorphism, SNP), in particular those potentially linked to resistance to anti-Pneumocystis treatments.

SECONDARY OUTCOMES:
to determine the factors associated (e.g. exposure to treatments) with P. jirovecii mutant strains | at inclusion

OTHER OUTCOMES:
to determine the impact of mutations on the effectiveness of anti-Pneumocystis treatment (e.g. favorable vs. unfavorable evolution of the infection) | 1 month and 3 month
to evaluate two methods - digital droplet PCR and biosensors without PCR - for the detection and characterization of mutations associated with resistance in Pneumocystis jirovecii | at inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement

REFERENCES:
- [Result] Hoffmann CV, Nevez G, Moal MC, Quinio D, Le Nan N, Papon N, Bouchara JP, Le Meur Y, Le Gal S. Selection of Pneumocystis jirovecii Inosine 5'-Monophosphate Dehydrogenase Mutants in Solid Organ Transplant Recipients: Implication of Mycophenolic Acid. J Fungi (Basel). 2021 Oct 10;7(10):849. doi: 10.3390/jof7100849. PMID 34682270
- [Result] Argy N, Le Gal S, Coppee R, Song Z, Vindrios W, Massias L, Kao WC, Hunte C, Yazdanpanah Y, Lucet JC, Houze S, Clain J, Nevez G. Pneumocystis Cytochrome b Mutants Associated With Atovaquone Prophylaxis Failure as the Cause of Pneumocystis Infection Outbreak Among Heart Transplant Recipients. Clin Infect Dis. 2018 Aug 31;67(6):913-919. doi: 10.1093/cid/ciy154. PMID 29514207
- [Result] Bonnet PL, Hoffmann CV, Le Nan N, Bellamy L, Hoarau G, Flori P, Demar M, Argy N, Morio F, Le Gal S, Nevez G. Atovaquone exposure and Pneumocystis jirovecii cytochrome b mutations: French data and review of the literature. Med Mycol. 2023 Sep 4;61(9):myad095. doi: 10.1093/mmy/myad095. PMID 37656874
- [Result] de la Horra C, Friaza V, Morilla R, Delgado J, Medrano FJ, Miller RF, de Armas Y, Calderon EJ. Update on Dihydropteroate Synthase (DHPS) Mutations in Pneumocystis jirovecii. J Fungi (Basel). 2021 Oct 13;7(10):856. doi: 10.3390/jof7100856. PMID 34682277
- [Result] Nahimana A, Rabodonirina M, Bille J, Francioli P, Hauser PM. Mutations of Pneumocystis jirovecii dihydrofolate reductase associated with failure of prophylaxis. Antimicrob Agents Chemother. 2004 Nov;48(11):4301-5. doi: 10.1128/AAC.48.11.4301-4305.2004. PMID 15504856
- [Result] Kojabad AA, Farzanehpour M, Galeh HEG, Dorostkar R, Jafarpour A, Bolandian M, Nodooshan MM. Droplet digital PCR of viral DNA/RNA, current progress, challenges, and future perspectives. J Med Virol. 2021 Jul;93(7):4182-4197. doi: 10.1002/jmv.26846. Epub 2021 Mar 11. PMID 33538349
- [Result] Pla L, Avino A, Eritja R, Ruiz-Gaitan A, Peman J, Friaza V, Calderon EJ, Aznar E, Martinez-Manez R, Santiago-Felipe S. Triplex Hybridization-Based Nanosystem for the Rapid Screening of Pneumocystis Pneumonia in Clinical Samples. J Fungi (Basel). 2020 Nov 17;6(4):292. doi: 10.3390/jof6040292. PMID 33213011